CLINICAL TRIAL: NCT04166812
Title: Role of Small Airway Dysfunction for Disease Progression in Early COPD - an Observational Two-year Study
Brief Title: Change in Airway Peripheral Tone in COPD
Acronym: CAPTO-COPD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Heidelberg University (Other)
Collaborators: PD Dr. Henrik Watz, Pulmonary Research Center, LungenClinic Großhansdorf (Principal Investigator) (Unknown); Chiesi GmbH, Hamburg, Germany (Funding) (Unknown)
Responsible Party: Principal Investigator, Dr. Frederik Trinkmann, Principial Investigator, Heidelberg University
Other Study IDs: CAPTO-COPD
Record Dates: First submitted 2019-11-12; First posted 2019-11-18 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: COPD; COPD, Early-Onset
Keywords: small airway disease; peripheral airway tone
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Spirometry; Plethysmography, Whole Body; Fractional Exhaled Nitric Oxide Testing; F Factor; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with early COPD: diagnosis according to current GOLD recommendations
  Interventions: Diagnostic Test: oscillometry; Diagnostic Test: multiple breath washout testing; Diagnostic Test: spirometry; Diagnostic Test: body plethysmography; Diagnostic Test: fractional exhaled nitric oxide; Diagnostic Test: transfer factor; Diagnostic Test: health status; Diagnostic Test: computed tomography; Diagnostic Test: induced sputum
- patients at risk for COPD: no current diagnosis according to GOLD recommendations, but at risk for COPD
  Interventions: Diagnostic Test: oscillometry; Diagnostic Test: multiple breath washout testing; Diagnostic Test: spirometry; Diagnostic Test: body plethysmography; Diagnostic Test: fractional exhaled nitric oxide; Diagnostic Test: transfer factor; Diagnostic Test: health status; Diagnostic Test: computed tomography; Diagnostic Test: induced sputum

INTERVENTIONS:
Diagnostic Test: oscillometry — assessment of peripheral airway resistance using oscillometry
Diagnostic Test: multiple breath washout testing — assessment of ventilation heterogeneity using multiple breath washout testing
Diagnostic Test: spirometry — assessment of lung function using spirometry
Diagnostic Test: body plethysmography — assessment of lung function using body plethysmography
Diagnostic Test: fractional exhaled nitric oxide — assessment of eosinophilic airway inflammation using fractional exhaled nitric oxide
Diagnostic Test: transfer factor — assessment of gas transfer using single breath transfer factor for carbon monoxide
Diagnostic Test: health status — assessment of health status using validated questionnaires (St. George's Respiratory Questionnaire [SGRQ], COPD Assessment Test [CAT])
Diagnostic Test: computed tomography — assessment of lung structure and function using computed tomography (only in patients with clinical indication, Heidelberg site)
Diagnostic Test: induced sputum — various biomarkers (subgroup of approximately 75 patients, Großhansdorf site)

SUMMARY:
Small airways disease is a pathological feature in mild to moderate COPD, which might be causally involved in disease progression. However, there are only limited studies available that prospectively identified patients at risk for small airway disease. Our intention is to investigate the early phase of the disease. In addition, we thereby want to build up a well-defined study population of patients in an early phase of the disease with a rapid decrease in lung function as measured by oscillometry and multiple breath washout (MBW)-testing. In addition, it is our goal to identify patients in an early stage of disease and patients at risk of fast progression and/or rapid decline in lung function.

ELIGIBILITY:
patients at risk for COPD

inclusion criteria:

* smoking history (at least 10 pack years)
* absence of airway obstruction (FEV1/FVC ≥ 70% after salbutamol 400µg)
* high symptom score (CAT ≥ 10) or long acting bronchodilator therapy
* age > 35 years

exclusion criteria:

* respiratory infection within 4 weeks prior to inclusion
* other symptomatic pulmonary disease, except bronchial asthma

patients with early COPD

inclusion criteria:

* smoking history (at least 10 pack years)
* mild COPD (FEV1/FVC < 70% and FEV1 ≥ 70% after salbutamol 400µg)
* age > 35 years

exclusion criteria:

* respiratory infection within 4 weeks prior to inclusion
* other pulmonary disease, except bronchial asthma

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * patients at risk for COPD with no current diagnosis according to GOLD recommendations
  * patients with early COPD with diagnosis according to current GOLD recommendations
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
oscillometry (change in R5-20) | 24 months
  change in frequency dependence of resistance (R5-20)
multiple breath washout testing (change in LCI) | 24 months
  change in global ventilation heterogeneity (lung clearance index, LCI)
multiple breath washout testing (change in Scond) | 24 months
  change in conductive ventilation heterogeneity (Scond)
multiple breath washout testing (change in Sacin) | 24 months
  change in acinar ventilation heterogeneity (Sacin)

SECONDARY OUTCOMES:
spirometry (change in FEV1) | 24 months
  change in parameters of central obstruction (forced expiratory volume in one second, FEV1)
body plethysmography (change in RV/TLC) | 24 months
  change in parameters of hyperinflation (residual volume / total lung capacity RV/TLC)
body plethysmography (change in sRaw) | 24 months
  change in specific airway resistance (sRaw)
health Status (change in SGRQ-c) | 24 months
  change in quality of life (SGRQ-c)
health Status (change in CAT) | 24 months
  change in symptom score (CAT)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Watz, MD, Principal Investigator — Pulmonary Research Institute at LungClinic Großhansdorf; Frederik Trinkmann, MD, Principal Investigator — Thoraxklinik at Heidelberg University
Locations (2):
- Germany (2):
  - Pulmonary Research Institute at LungClinic Großhansdorf, Großhansdorf
  - Thoraxklinik at Heidelberg University, Heidelberg

IPD SHARING:
Plan to Share IPD: No
data protection rules do not allow to share individual participant data